CLINICAL TRIAL: NCT03105401
Title: Phenomenological and Psychopathological Factors Associated to Hallucinations in Parkinson's Disease
Acronym: HALLUPARK
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulties
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0137
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients affected by Parkinson's disease: Outpatients affected by Parkinson's Disease consulting in neurology can be included if volunteer
  Interventions: Other: Assessment of hallucinations in Parkinson's disease

INTERVENTIONS:
Other: Assessment of hallucinations in Parkinson's disease — Patients participating to the study will be asked to answer a semi-structured questionnaire searching for hallucinations of all modalities, minor psychotic symptoms and delusions. Psychometric scales will be assessed to search for depressive symptoms, cognitive impairment and specific personality characteristics.

SUMMARY:
This study aims to describe hallucinations prevalence in a sample of patients affected by Parkinson's disease and consulting in an outpatient facility.

An unique one hour interview will be offered to volunteers patients. Patients participating to the study will be asked to answer a semi-structured questionnaire searching for hallucinations of all modalities, minor psychotic symptoms and delusions. Psychometric scales will be assessed to search for depressive symptoms, cognitive impairment and specific personality characteristics.

The study hypothesis is that hallucinations prevalence in Parkinson's disease is underestimated and is higher than usually described in the scientific literature when all hallucinations modalities and minor hallucinatory phenomenons are searched for.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years-old
* Absence of opposition from the patient himself/herself or his/her legal representant for his/her participation to the study
* Patient without superior age limit with a diagnosis of Parkinson's disease made according to the UKPDSBB criteria (UK Parkinson's Disease Society Brain Bank clinical diagnostic criteria)
* Outpatient consulting in neurology at the Charpennes'hospital

Exclusion Criteria:

* Opposition to the study
* Deafness or blindness which could compromise the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients affected by Parkinson's Disease consulting in neurology can be included if volunteer
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Hallucinations Prevalence | 1 hour
  Semi-structured questionnaire precisely describing hallucinations of all modalities and their characteristics, as well as minor hallucinations and delusions. Binary Yes/No possible answers.
  Unique 1 hour interview to assess semi-structured questionnaire for primary outcome measurement, and psychometric scales.

CONTACTS AND LOCATIONS:
Overall Officials: Jing XIE, MD, Principal Investigator — Hôpital des Charpennes. Centre de Recherche Clinique - vieillissement, cerveau, fragilité
Locations (1):
- Hôpital des Charpennes. Centre de Recherche Clinique - vieillissement, cerveau, fragilité, Villeurbanne, France